CLINICAL TRIAL: NCT06369766
Title: Retinal Markers in Neuroinflammatory Diseases: a Prospective Observational Study
Brief Title: REtinal Markers In Neuroinflammatory Diseases ("REMIND")
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02144; ko23Papadopoulou4
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Neuroinflammatory Diseases
Keywords: Retinal Markers; OCT; Disease Progression; Progression Independent of Relapse Activity (PIRA)
MeSH Terms: conditions — Multiple Sclerosis; Neuroinflammatory Diseases; Disease Progression | interventions — Tomography, Optical Coherence; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: Healthy control subjects without neurological diseases
  Interventions: Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Static retinal vessel analyzer; Diagnostic Test: Dynamic retinal vessel analyzer; Diagnostic Test: Laser speckle flowgraphy system; Other: Questionnaire
- Patients with Multiple Sclerosis
  Interventions: Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Static retinal vessel analyzer; Diagnostic Test: Dynamic retinal vessel analyzer; Diagnostic Test: Laser speckle flowgraphy system; Other: Questionnaire
- Patients with other neuroinflammatory diseases of the CNS
  Interventions: Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Static retinal vessel analyzer; Diagnostic Test: Dynamic retinal vessel analyzer; Diagnostic Test: Laser speckle flowgraphy system; Other: Questionnaire

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography (OCT) — OCT is used to measure:
  * peripapillary retinal nerve fiber layer (mean thickness in μm)
  * ganglion cell-inner plexiform layer (volume in mm^3 and mean thickness in μm)
  * other retinal layers (inner nuclear layer, outer plexiform layer, outer nerve layer; volumes in mm^3 and mean thickness in μm).
  The "scanner laser ophthalmoscopy"-function of the OCT device is used to continuously record the exact location of each participant's fixation point in relation to their fovea and thereby allows the assessment of the fixation instability.
  In a subgroup of participants, the "angiography"-module of the OCT device is used to image the retinal blood flow and thereby allows to measure the vascular area density of the superficial retinal capillary plexus and deep retinal capillary plexus.
Diagnostic Test: Static retinal vessel analyzer — Static retinal vessel analyzer is used to determine:
  * central retinal arteriolar diameter equivalents (in μm)
  * central retinal venular diameter equivalents (in μm)
  * arteriolar-to-venular diameter ratio
Diagnostic Test: Dynamic retinal vessel analyzer — In a subgroup of participants, the dynamic retinal vessel analyzer is used to determine the arteriolar ficker light-induced dilatation, venular ficker light-induced dilatation, and Arteriolar constriction, measured in % dilatation in comparison to baseline.
Diagnostic Test: Laser speckle flowgraphy system — In a subgroup of participants, the laser speckle flowgraphy system is used to measure the relative ocular blood flow as expressed in arbitary units of Mean Blur Rate.
Other: Questionnaire — All study participants will be asked to fill in a questionnaire with various questions regarding existing eye diseases, other diseases (including vascular diseases/risk factors), and daily physical activity that could influence the results of the retinal examinations. Physical activity will be assessed using an adapted form of the standardized Global Physical Activity Questionnaire.

SUMMARY:
The goal of this observational study, including patients with Multiple Sclerosis, patients with other neuroinflammatory diseases and healthy controls, is to determine the predictive value of retinal markers in predicting disease progression. Participants complete a questionnaire and undergo various non-invasive retinal routine clinical examinations.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an autoimmune disease of the central nervous system (CNS) and represents one of the most common neurological disorders affecting young adults worldwide and often leads to significant disability over time. While MS typically presents with recurrent neurological symptoms known as relapses, most patients also experience progressive neurological deterioration independent of relapses, referred to as progression independent of relapse activity (PIRA). PIRA is a major contributor to long-term disability and represents a significant challenge in the management of MS. Early identification of patients at high risk to develop PIRA is crucial for therapeutic decisions and testing treatment efficacy, highlighting the urgent need for accurate predictive markers of progression in MS.

The primary objective of this longitudinal, observational, prospective, single center study is to investigate the predictive value of various retinal markers in predicting PIRA in MS patients.

The study assesses several easily obtained, non-invasive retinal measures:

* Neuroaxonal loss in the retina: This serves as a marker of neurodegeneration in the CNS. It will be assessed by measuring the volume of the ganglion cell-inner plexiform layer and the thickness of the peripapillary retinal nerve fiber layer using optical coherence tomography (OCT).
* Neuroinflammation in the retina: This will be assessed by evaluating thickening of other retinal layers in OCT, particularly the inner nuclear layer.
* Fixation instability of the patients: This serves as a marker of global neuronal dysfunction in the CNS. It will be measured using Scanner Laser Ophthalmoscopy-OCT.
* Structural changes of the retinal vessels: Particularly, the arteriolar and venular diameters will be assessed. This serves as a marker of systemic microvascular health and will be measured using static retinal vessel analysis.
* Functional/perfusional changes of the retinal vessels: For a subgroup of patients, this will be evaluated using OCT-angiography, and/or dynamic retinal vessel analysis, and/or laser speckle flowgraphy. These measures provide insights into the functional and perfusional changes of the retinal vessels.

As secondary objectives, this study comprises:

* Comparison with other biomarkers of neuroaxonal damage to determine whether the retinal markers are independent and/or stronger predictors of PIRA.
* Comparison with the retinal markers of Healthy Controls and patients with other neuroinflammatory diseases of the CNS to understand the differences in mechanisms of damage.
* Investigating the associations among the various retinal measures to understand the relationship between neuroaxonal loss, functional deficits and vascular changes in MS.

Data will be collected at baseline and annually over up to 5 years, or for some MS patients, up to 10 years, to evaluate changes in retinal markers and their correlation with disease progression. This comprehensive assessment will provide valuable insights into the utility of retinal markers in predicting PIRA and their relationship with disease severity and progression in MS.

ELIGIBILITY:
Inclusion Criteria:

1. All groups:

   * Age >18 years old
2. Patients with Multiple Sclerosis:

   * Diagnosis of Multiple Sclerosis, according to the last revisions of the McDonald Criteria (2017)
3. Patients with other neuroinflammatory diseases:

   * Diagnosis of Neuromyelitis optica spectrum disorder or Myelin oligodendrocyte glycoprotein antibody disease or other neuroinflammatory disorders other than Multiple Sclerosis

Exclusion Criteria:

1. All groups:

   * Inability to undergo Optical Coherence Tomography (OCT) and/or retinal vessel imaging (e.g. severe nystagmus that prevents eye fixation on both eyes)
   * Presence of any ocular pathology that may interfere with the validity of the OCT/retinal vessel analysis (cataracts, glaucoma, history of refractive defects >6 D etc.).
   * Pregnancy and Lactation
2. Healthy Controls

   * History of other neurological conditions: participants with a history of other significant neurological conditions that might interfere with the assessment or interpretation of the signs and symptoms will be excluded (e.g. confirmed Stroke, Acute disseminated encephalomyelitis, Chronic inflammatory Demyelinating Disease, Polyneuropathy, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis and the other neuroinflammatory diseases are recruited in the Multiple Sclerosis and Neuroimmunology center of the Department of Neurology at the University Hospital Basel in Basel. These patients with Multiple Sclerosis are participants of the ongoing observational Swiss Multiple Sclerosis Cohort Study. Healthy Controls are recruited from an older healthy control-cohort, which were matched to the Multiple Sclerosis patients and underwent Optical Coherence Tomography in 2016/2017. Further Healthy Controls are recruited bycontacting volunteers that participated in previous studies and agreed to be contacted again for new studies and by public announcements.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Occurence of Progression Independent of Relapse Activity (PIRA) | 5 Years (or for a subgroup up to 10 years) after baseline
  The group of "Multiple Sclerosis patients" undergo a detailed neurological interview and examination for the calculation of the Expanded Disability Status Scale (EDSS) at each clinical visit every 6 or 12 months. The EDSS worsening is used to define PIRA retrospectively (increase of ≥1.5 points if baseline EDSS was 0 points, increase of ≥1.0 points if baseline EDSS was 1-5.5 points or increase of ≥0.5 point if baseline EDSS was >5.5 points), with no relapse between the reference- event- and confirmation score visits. Relapse is defined as objectively observed signs typical of an acute CNS inflammatory demyelinating event, with duration of at least 24hours in the absence of fever or infection, separated from the last relapse by ≥30 days. The occurence of PIRA (yes/no) is assessed at the end of the follow-up period of the different retinal markers (5 years or for a subgroup up to 10 years after baseline).
Neuroaxonal loss in the retina (as marker of neurodegeneration in the CNS) | Baseline and once every year over up to 5 years
  To determine the neuroaxonal loss in the retina, the thickness of the peripapillary retinal nerve fiber layer and the volume of the ganglion cell-inner plexiform layer are assessed by optical coherence tomography (OCT).
Neuroinflammation in the retina | Baseline and once every year over up to 5 years
  To determine the neuroinflammation in the retina, the thickening of the outer plexiform layer, outer nerve layer and ,in particular, of the inner nuclear layer are assessed by OCT.
Fixation instability (as marker of global neuronal dysfunction in the CNS) | Baseline and once every year over up to 5 years
  To determine the fixation instability, visual fixation measurements are recorded via the "Scanner Laser Ophthalmoscopy"-function of the OCT device (as described by Mallery et al., 2018; PMID: 29340646).
Structural changes of the retinal vessels (as marker of systemic microvascular health) | Baseline and once every year over up to 5 years
  To determine structural changes of the retinal vessels, the retinal arterior and venular diameters are measured by static retinal vessel analysis.
(For a subgroup of participants) Functional/perfusional changes of the retinal vessels | Baseline and once every year over up to 5 years
  To determine the functional/perfusional changes of the retinal vessels, a subgroup of participants (patients= 100, Healthy Controls= 50) undergoes additional examinations:
  * OCT-Angiography: measurement of retinal perfusion
  * Dynamic Retinal vessel analysis: measurement examining the motility and function of the retinal vessels
  * Laser Speckle Flowgraphy: measurement of ocular perfusion

SECONDARY OUTCOMES:
Relative value of retinal markers for the prediction of PIRA compared to or combined with other biomarkers of neuroaxonal damage | Baseline and once every year over up to 5 years
  Data regarding other biomarkers (serum neurofilament light chain and brain volume on magnet resonance imaging) that are already available within the clinical routine and/or the SMSC study are used to assess the relative value of the retinal markers described above under primary outcome measures 2-6 in predicting PIRA, both independently or in combination with these other biomarkers.
Comparison of the examined retinal markers of Multiple Sclerosis patients with Healthy Controls and with patients with other neuroinflammatory diseases of the CNS | Baseline and once every year over up to 5 years
  Examined retinal markers are compared between the different groups to understand the relationship among the different measures independently of disease.
The relationship between neuroaxonal loss, functional deficits and vascular changes in Multiple Sclerosis | Baseline and once every year over up to 5 years
  Investigation of the associations among the examined retinal measures to understand the relationship between neuroaxonal loss, functional deficits and vascular changes in Multiple Sclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Athina Papadopoulou, PD Dr. med., Principal Investigator — University Hospital Basel, Department of Neurology
Locations (1):
- University Hospital Basel, Department of Neurology, Basel, Switzerland